CLINICAL TRIAL: NCT02202720
Title: Evaluation of Richmond Agitation Sedation Scale According to Alveolar Concentration of Sevoflurane During a Sedation With Sevoflurane in ICU Patients
Acronym: SEVORASS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0200; 2014-000759-10
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Requiring Sedation by Sevoflurane in ICU; Adult Patients; Patients Covered by French Health Care System; Patients Who Have Given Their Consent
Keywords: Sevoflurane; RASS score; Sedation; Minimal alveolar concentration (MAC)
MeSH Terms: interventions — Sevoflurane

ARMS (1):
- sevoflurane (Experimental)
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — Short term sedation with sevoflurane in ICU

SUMMARY:
Describe the Richmond Agitation Sedation Scale (RASS) values corresponding to the values of Minimum alveolar concentration of sevoflurane during sedation of patients in ICU

DETAILED DESCRIPTION:
Prospective clinical study in ICU with sedated ventilated patients with sevoflurane using the Mirus® system. Pharmacological study of the concentration-effect relationship by administration at increasing and decreasing concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Requiring sedation by sevoflurane in ICU
* Adult patients
* Patients covered by french health care system
* Patients who have given their consent or his family

Exclusion Criteria:

* Pregnant or lactating women
* Sevoflurane anaphylaxia
* Known or suspected risk of malignant hyperthermia
* Refusal Protocol
* Brain-damaged patients
* Hemodynamic conditions not compatible with the use of sevoflurane
* ARDS patients
* Minor patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Description of the RASS score | at day 1
  Describe the RASS score corresponding to the values of sevoflurane MAC during sedation of patients in ICU : RASS score determined at the middle of each level of 30 minutes, each level correspond to determined sevoflurane MAC with ascending MAC ranging from 0 to 0.8 and then descending MAC from 0.8 to 0.

SECONDARY OUTCOMES:
determination of the associated hemodynamic and respiratory parameters | at day 1
  Determine the associated hemodynamic and respiratory parameters, bispectral index and analgesia-nociception index for each level of sevoflurane MAC (monitored at the middle of each level of 30 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France